CLINICAL TRIAL: NCT02646150
Title: Clinical Use of Magnetic Resonance Perfusion Imaging to Qualitatively Assess Adequate Distal Perfusion After Endovascular Revascularization in Critical Limb Ischemia
Acronym: MR CLI
Status: Completed | Type: Observational
Sponsor: Seung-Whan Lee, M.D., Ph.D. (Other)
Responsible Party: Sponsor-Investigator, Seung-Whan Lee, M.D., Ph.D., Division of Cardiology, Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: AMCCV2015-10
Record Dates: First submitted 2016-01-04; First posted 2016-01-05 (Estimated); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Lower Limb; Ischemia; Perfusion
Keywords: Magnetic Resonance perfusion imaging; distal perfusion; Critical Limb Ischemia; endovascular revascularization
MeSH Terms: conditions — Ischemia; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- critical limb ischemia
  Interventions: Procedure: Magnetic Resonance Perfusion Imaging

INTERVENTIONS:
Procedure: Magnetic Resonance Perfusion Imaging

SUMMARY:
This study evaluates the clinical effectiveness of Magnetic Resonance(MR) perfusion imaging to qualitatively assess adequate distal perfusion after endovascular revascularization in Critical Limb Ischemia

ELIGIBILITY:
Inclusion Criteria:

* Age 20 and above
* Critical limb ischemia with ulcer
* Ankle brachial index(ABI) ≤ 0.9 or Toe brachial index (TBI) ≤ 0.5 or Transcutaneous oxygen pressure (TcPo2) ≤ 40mmHg
* ≥ 70 percentage of stenosis of infrapopliteal artery on lower extremity computed tomography angiography or lower extremity doppler
* Subject understands protocol and provides written, informed consent

Exclusion Criteria:

* Post-traumatic critical limb ischemia
* Neurogenic limb ischemia
* Life expectancy ≤ 2 years

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lower extremity ischemia
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2015-12-12 (Actual); Primary Completion 2021-07-13 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
The change of deoxyhemoglobin in MR imaging | 6 months

SECONDARY OUTCOMES:
The event rate of unplanned major and minor amputation in limb | 6 months
The event rate of complete healing of lower extremity ulcer | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
This trial is not publicly funded clinical trial.